CLINICAL TRIAL: NCT06570642
Title: Using Real-Time Data Capture to Examine Affective Mechanisms as Mediators of Physical Activity Adherence in Interventions
Brief Title: eMOTION: Examining Affective Mechanisms in Physical Activity Engagement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Genevieve Dunton, Chief, Division of Health Behavior Research and Director, USC Real-Time Eating Activity and Children's Health (REACH) Lab, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: UP-22-00332; R01CA272933 (NIH)
Record Dates: First submitted 2024-08-16; First posted 2024-08-26 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Physical Inactivity; Overweight or Obesity; Cancer
Keywords: Affective Response; Psychological Needs; Physical Activity
MeSH Terms: conditions — Sedentary Behavior; Overweight; Obesity; Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study will use a partial factorial, crossover, within x between subjects design. Participants randomly receive affect- or intensity-based goals for 8-weeks (Part 1), followed by a 2-week washout period, then cross-over to the other condition for 8-weeks (Part 2). During the affect-based goal condition, participants randomly receive one of four combinations of intervention enhancements: TYPE/CONTEXT (with vs. without) x SAVOR (with vs. without). In summary, participants are randomly assigned to one of eight groups based on order and intervention components: (1) intensity > affect without enhancements; (2) intensity > affect with TYPE/CONTEXT; (3) intensity > affect with SAVOR; (4) intensity > affect with both TYPE/CONTEXT and SAVOR; (5) affect without enhancements > intensity; (6) affect with TYPE/CONTEXT > intensity; (7) affect with SAVOR > intensity; and (8) affect with both TYPE/CONTEXT and SAVOR > intensity.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Affect (no enhancements) > Intensity (Experimental): Participants receive affect-based goals for the first 8-weeks, then cross-over to receive intensity-based goals for the second 8-weeks. No enhancements are added to the standard mHealth intervention.
  Interventions: Behavioral: Physical Activity Goals mHealth Intervention
- Intensity > Affect (no enhancements) (Experimental): Participants receive intensity-based goals for the first 8-weeks, then cross-over to receive affect-based goals for the second 8-weeks. No enhancements are added to the standard mHealth intervention.
  Interventions: Behavioral: Physical Activity Goals mHealth Intervention
- Affect (+ SAVOR + TYPE/CONTEXT) > Intensity (Active Comparator): Participants receive affect-based goals for the first 8-weeks. In addition to the standard mHealth intervention, participants engage in both SAVOR and TYPE/CONTEXT enhancements to augment the treatment effects of the affect-based goals condition. Participants then cross-over to receive intensity-based goals for the second 8-weeks.
  Interventions: Behavioral: Physical Activity Goals mHealth Intervention; Behavioral: TYPE/CONTEXT enhancement; Behavioral: SAVOR enhancement
- Intensity > Affect (+ SAVOR + TYPE/CONTEXT) (Active Comparator): Participants receive intensity-based goals for the first 8-weeks, then cross-over to receive affect-based goals for the second 8-weeks. In addition to the standard mHealth intervention, participants engage in both SAVOR and TYPE/CONTEXT enhancements to augment the treatment effects of the affect-based goals condition.
  Interventions: Behavioral: Physical Activity Goals mHealth Intervention; Behavioral: TYPE/CONTEXT enhancement; Behavioral: SAVOR enhancement
- Affect (+SAVOR) > Intensity (Active Comparator): Participants receive affect-based goals for the first 8-weeks. In addition to the standard mHealth intervention, participants engage in the SAVOR enhancement to augment the treatment effects of the affect-based goals condition. Participants then cross-over to receive intensity-based goals for the second 8-weeks.
  Interventions: Behavioral: Physical Activity Goals mHealth Intervention; Behavioral: SAVOR enhancement
- Intensity > Affect (+SAVOR) (Active Comparator): Participants receive intensity-based goals for the first 8-weeks, then cross-over to receive affect-based goals for the second 8-weeks. In addition to the standard mHealth intervention, participants engage in the SAVOR enhancement to augment the treatment effects of the affect-based goals condition.
  Interventions: Behavioral: Physical Activity Goals mHealth Intervention; Behavioral: SAVOR enhancement
- Affect (+TYPE/CONTEXT) > Intensity (Active Comparator): Participants receive affect-based goals for the first 8-weeks. In addition to the standard mHealth intervention, participants engage in the TYPE/CONTEXT enhancement to augment the treatment effects of the affect-based goals condition. Participants then cross-over to receive intensity-based goals for the second 8-weeks.
  Interventions: Behavioral: Physical Activity Goals mHealth Intervention; Behavioral: TYPE/CONTEXT enhancement
- Intensity > Affect (+TYPE/CONTEXT) (Active Comparator): Participants receive intensity-based goals for the first 8-weeks, then cross-over to receive affect-based goals for the second 8-weeks. In addition to the standard mHealth intervention, participants engage in the TYPE/CONTEXT enhancement to augment the treatment effects of the affect-based goals condition.
  Interventions: Behavioral: Physical Activity Goals mHealth Intervention; Behavioral: TYPE/CONTEXT enhancement

INTERVENTIONS:
Behavioral: Physical Activity Goals mHealth Intervention — On days participants plan to exercise, they engage in two daily goal sessions (morning and evening). Morning sessions provide an activity goal for the day and ask the participant to create a plan, anticipate barriers, and brainstorm solutions for achieving this goal. The affect-based goal condition asks participants to engage in either (1) a type (50% of daily goals) or (2) a context (50% of daily goals) of physical activity that allows them to experience positive affect. Goals focused on context are randomly generated to suggest that the participant performs activity (1) in a place; (2) in a social situation; or (3) while listening to something that makes them feel good. The intensity-based goal condition asks participants to maintain a certain target heart rate range during physical activity. Starting heart rate reflects the approximate age-adjusted heart rate max, with goals progressively increasing from 55% to 70% heart rate max.
Behavioral: TYPE/CONTEXT enhancement — TYPE/CONTEXT augments intervention effects by providing tailored recommendations for activity types and contexts that satisfy personally-important psychological needs as rated by each participant at baseline. Ratings from a crowdsourced panel of adults on Amazon Mechanical Turk will be used to determine the potential for specific activity types and contexts to satisfy psychological needs; our tailoring algorithm will then recommend the corresponding activity type or context while accounting for reported constraints (e.g., ability, access). These details will be incorporated into a tailored recommendation provided to participants each Sunday as they make activity plans for the upcoming week. Specifically, the program will randomly select either type or context (i.e., location, audio, social) recommendations and will rotate every two weeks. For TYPE, participants' top 3 activity types are recommended; for CONTEXT, participants' top 3 activity contexts are recommended.
  Arms: Affect (+ SAVOR + TYPE/CONTEXT) > Intensity; Affect (+TYPE/CONTEXT) > Intensity; Intensity > Affect (+ SAVOR + TYPE/CONTEXT); Intensity > Affect (+TYPE/CONTEXT)
Behavioral: SAVOR enhancement — SAVOR implements a brief savoring exercise on the smartphone that takes place either after the planned physical activity session or during the evening goal session (after the self-monitoring module). Participants will respond to questions that are intended to enhance and prolong positive experiences during physical activity. To trigger attentional deployment, a common savoring strategy that involves intensifying experiences by focusing on them, participants will answer three open-ended prompts. These prompts are drawn from a prompt pool with slightly varied wording to promote a sense of novelty. Savoring prompts will rotate daily and have a day lag built in every week (i.e., Week 1 Monday Savoring Prompts are Week 2 Tuesday Savoring Prompts).
  Arms: Affect (+ SAVOR + TYPE/CONTEXT) > Intensity; Affect (+SAVOR) > Intensity; Intensity > Affect (+ SAVOR + TYPE/CONTEXT); Intensity > Affect (+SAVOR)

SUMMARY:
This early-phase trial will test intervention strategies to influence affective mechanisms underlying physical activity and determine whether changes in those mechanisms result in change in physical activity behavior among inactive adults who are overweight or obese.

DETAILED DESCRIPTION:
This ORBIT model phase 1 trial will examine whether affective mechanisms (1) can be experimentally manipulated in real-world settings; and (2) mediate the relationship between interventions and physical activity behavior. A novel physical activity intervention will be optimized by efficiently disentangling the effects of its core component and two enhancement components on affective mechanisms associated with physical activity engagement.

ELIGIBILITY:
Inclusion criteria:

1. Aged ≥ 18 years
2. Reside in the United States
3. Self-reported BMI ≥ 25
4. Current structured physical activity engagement < 60 minutes per week
5. Own a personal smartphone device
6. Reside in an area with Internet or Wi-Fi connectivity during the study period
7. Able to speak and read in English
8. Interested and willing to start a physical activity program
9. Willing to wear a Fitbit Versa smartwatch provided by the study team everyday continuously (including at work and during physical activity), in place of any Fitbits or smartwatches previously worn, for the duration of the study period
10. Able to read the small font on a smartwatch screen without glasses, or willing to carry reading glasses during physical activity for the purpose of reading the smartwatch screen

Exclusion Criteria:

1. Inability to provide informed consent due to cognitive disability
2. Inability to engage in one or more key treatment components, including those with medical conditions that preclude physical activity engagement or who cannot wear an accelerometer on the wrist or answer brief surveys on the smartwatch for any reason
3. Current pregnancy
4. Referred to the study by another participant or from Reddit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Physical Activity: Step Count | Daily total for weeks 1-19
  Daily steps will be calculated from minute-level accelerometer data. Fitbit Versa 3 smartwatches with internal accelerometers are worn for the duration of the study period, except while bathing or charging. Only days with sufficient wear time (defined as ≥ 10-hours of valid data, where no more than 20-minutes per hour has a consecutive step count of zero) are used for analysis.
Physical Activity: Minutes | Daily total for weeks 1-19
  Daily minutes of light, moderate, and vigorous physical activity will be calculated from minute-level accelerometer data. Fitbit Versa 3 smartwatches with internal accelerometers are worn for the duration of the study period, except while bathing or charging. Only days with sufficient wear time (defined as ≥ 10-hours of valid data, where no more than 20-minutes per hour has a consecutive step count of zero) are used for analysis.

SECONDARY OUTCOMES:
Affective Response | Max 2 per 60-min physical activity period during weeks 2-9 and weeks 12-19
  Event-contingent ecological momentary assessment (EMA) check-ins sent to the smartwatch during physical activity measure affective response. Event-contingent EMA are triggered when Fitbit sensors detect physical activity via moving average heart rate. A ≥30-minute buffer separates the first and second EMA during a single physical activity bout. A maximum of two event-contingent EMA will be sent within any given 60-minute period. Participants are asked to safely pause their activity to answer seven items about their affective response using a 5-point bipolar Likert Scale. Five items (Energetic-Fatigued, Happy-Discouraged, Relaxed-Tense, Excited-Bored, Satisfied-Frustrated) are drawn from Russell's Circumplex Model of Affect; one (Good-Bad) represents core affective valence; and one (Proud-Embarrassed) represents self-conscious emotion.
Affectively-Charged Motivations | Up to once daily for weeks 2-9 and weeks 12-19
  Affectively-charged motivations for physical activity are measured during the morning goal session via REDCap. A text message alerts participants to complete the morning goal session on their smartphone. A single item from the Attraction-Antipathy subscale of the AFFEXX measures affectively-charged motivation by asking, "How do you feel about doing physical activity today?". Participants select a response using a Visual Analogue Scale ranging from 0 (Dread) to 100 (Excited).
Anticipated Affect | Up to once daily for weeks 2-9 and weeks 12-19
  Anticipated affect is measured during the morning goal session via REDCap. A text message alerts participants to complete the morning goal session on their smartphone. A single item asks, "How do you expect to feel during physical activity today?". Participants select a response using a Visual Analogue Scale ranging from 0 (Miserable) to 100 (Thrilled).

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve F Dunton, PhD MPH, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dunton GF, Hatzinger L, Crosley-Lyons R, Hewus M, Wang WL, Van Dyck D, Huh J. Randomized trial of a digital therapeutics intervention to enhance affective response during physical activity: Protocol for the eMOTION study. Contemp Clin Trials. 2025 Jul;154:107945. doi: 10.1016/j.cct.2025.107945. Epub 2025 May 12. PMID 40368026